CLINICAL TRIAL: NCT04671264
Title: Efficacy and Safety of Vibrating Capsule in the Treatment of Functional Constipation: a Multicenter, Double-blind, Randomized, Placebo-controlled Clinical Study
Brief Title: Efficacy and Safety of Vibrating Capsule in Patients With Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Changhai Hospital, Naval Medical University, Shanghai, China. (Unknown); Beijing Xiehe Hospital, Beijing 100000, China. (Unknown); Beijing Jishuitan Hospital, Beijing 100009, China. (Unknown); Tianjin Medical University General Hospital (Other); Qilu Hospital of Shandong University (Other); Zhejiang Province Hospital of TCM, The First Affiliated Hospital of Zhejiang TCM University, Hangzhou, China. (Unknown)
Responsible Party: Principal Investigator, Zhuan Liao, Principal Investigator, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vibrating Capsule II
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Functional Constipation; Gastrointestinal Disease; Capsule Endoscopy
Keywords: Vibrating capsule; Functional Constipation; Spontaneous Bowel Movement; Clinical Trial
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VC group (Experimental): Vibrating capsule (VC) was proposed and applied for the patent by professor Liao Zhuan from Changhai Hospital, developed and manufactured by the Ankon Medical Technology Co., Ltd. The system consisted of a vibrating capsule and an external configuration device (ECD). It's 26.7 mm in length, 11.8 mm in diameter and 4.5 + 0.5 g in weight.
  Each VC has its own semiconductor chip with serial number in order to be recognized and controlled by ECD. VC can be stopped by ECD or mobile-phone application. There was a bidirectional radio frequency communication signal between VC and ECD. In addition, an application (APP) named VCP can be connected to ECD through smart phone to select mode and debug specific parameters for VC. The capsule can be activated by ECD, and then the vibration mode can be controlled by a configurator or an smartphone application.
  Interventions: Device: Sallowing VC during six weeks
- Control group (Placebo Comparator): The Intervention of control group were similar to VC group except the capsule function. Sham capsule we used in control group which had no function of vibrating.
  Interventions: Device: Sallowing VC during six weeks

INTERVENTIONS:
Device: Sallowing VC during six weeks — follow-up was required for at least 6 times, once every two weeks through the whole study.
  For patients who had no colonoscopy examination within a year, colonoscopy was a must to exclude organic diseases.
  These included blood routine, blood biochemistry, urine routine, fecal routine, fecal occult blood, thyroid stimulating hormone (TSH), blood pregnancy test and ECG examination. Patients should finish all the examination in the run-in period and at the end of treatment period.
  Dairy cards were designed mainly for the record of the daily defecation of patients and filled out by the enrolled patients, and the content included date, whether the patients swallow capsules (time), whether the patients discharge capsules (time), defecation, defecation time, degree of defecation exertion(0~4), BSF scale, complete or incomplete defecation, whether the patient had the sense of anal obstruction, whether manual assistance was applied, and whether first-aid medicine was used (bisacodyl).
  Other Names: Performing and reporting colonoscopy; Having laboratory examination; Filling diary cards; Evaluating the satisfaction

SUMMARY:
The safety and efficacy of vibrating capsule (VC) in promoting defecation by mechanical stimulation of the gastrointestinal walls have been elucidated in animal studies and pilot clinical studies. Our study aimed to explore the clinical application of a newly developed smartphone-controlled multi-mode VC in the treatment of functional constipation (FC) on multicentres.

Patients referred to gastroenterology outpatient of Changhai Hospital with FC and met the eligible criteria for more than 6 months and with spontaneous complete bowel movement (SCBM) less than 3 times per week within recent 3 weeks were eligible for this study. The study was discussed with patients who satisfied the enrolment criteria and provided written informed consents.

DETAILED DESCRIPTION:
This study was a multicentred, double-blind, placebo-controlled clinical trial to assess the safety and the effecacy of a newly developed gastrointestinal vibrating capsule (VC) in treating patients with functional constipation (FC). The whole process included two weeks run-in period, six weeks double-blind, placebo-controlled treatment period, and a follow-up period until the discharge of all swallowed capsules. During treatment period, patients were required to swallow one capsule every three to four days and a total of twelve capsules.

For each patient, a face to face follow-up was required for at least 6 times, once every two weeks through the whole study.

Run-in period (Visit 1) Face to face consultation in gastroenterology outpatient clinic and sign of written informed consents; Barium enema or colonoscopy (no re-examination is needed if the patient has undergone barium enema or total colonoscopy within a year); Distribution of bisacodyl tablets and diary cards; Perform the following examinations: vital signs, physical examination and laboratory examination; Eligibility evaluation based on the entry/discharge criteria; Record of past medical history, concomitant diseases and medication; Collection of the baseline characteristics of the enrolled patients including age, sex, duration of constipation, mean SCBMs, spontaneous bowel movements (SBMs), BMs, frequency of bisacodyl tablets taken and Bristol Score.

Treatment period Visit 2： Randomization; Patients were asked to fill in PAC-SYM, PAC-QOL and Comprehensive Evaluation Questionnaire; Record of vital signs and physical examination; Distribution of bisacodyl tablets, capsule retrieving bags and VCs; Instruct patients how to use the control board and start the vibration of VCs; Recycle of bisacodine tablets; Distribution and collection of diary cards; Record of adverse events, concomitant diseases and medication. Visit 3, Visit 4： Patients were asked to fill in PAC-SYM, PAC-QOL and Comprehensive Evaluation Questionnaire; Record of vital signs and physical examination; Recheck fecal routine and occult blood examination; Distribution of bisacodyl tablets, capsule retrieving bags and VCs; Recycle of bisacodyl tablets and VCs; Distribution and collection of diary cards; Record of adverse events, concomitant diseases and medication. Visit 5： Patients were asked to fill in PAC-SYM, PAC-QOL and Comprehensive Evaluation Questionnaire; Record of vital signs and physical examination; ECG; Blood routine/blood biochemistry/urine routine; Fecal routine and occult blood; Recycle of bisacodyl tablets and VCs; Distribution and collection of diary cards; Distribution of capsule retrieving bags; Record of adverse events, concomitant diseases and medication.

Follow-up period (Visit6):

Determine the discharge of all capsules; Recycle of capsules; Collection of diary cards; During the follow-up period, once the capsule was discharged the follow-up would be ended. If the capsules were still in the body, the patients must continue the follow-up until the capsules were all discharged.

The primary endpoint was the proportion of patients with SBM increased more than 1 time during treatment period. Secondary endpoints including mean SCBM , SBM , bowel movement (BM) and their improvements , Bristol Score, capsule evacuation time and satisfaction level. Patients were continuously monitored for adverse events (AE) at baseline and at each visit. Satisfaction level were evaluated based on Patient Assessment of Constipation Quality of Life questionnaire (PAC-QOL) and Patient Assessment of Constipation Symptom (PAC-SYM) at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged over 18 years and under 80 years;
* Patients who present with chronic constipation for more than 6 months and with SBM less than 3 times per week within recent 3 weeks and have at least one of the following symptoms for more than one-fourth (25%) during defecation:

  1. Straining;
  2. Lumpy or hard stools (bristol stool form (BSF scale 1~2);
  3. Sensation of incomplete evacuation;
  4. Sensation of anorectal obstruction/blockage;
  5. Manual maneuvers to facilitate defecation. Note: The above criteria can only be applied during spontaneous defecation, including no taking of laxatives within 24 hours before defecation, etc.
* Organic diseases were not found by barium enema or colonoscopy in the past year.
* Insufficient criteria for irritable bowel syndrome.

Exclusion Criteria:

* Patients who have contraindications to gastroscopy or colonoscopy;
* Patients under 18 years or over 80 years;
* Active vomiting;
* Patients with a permanent pacemaker (e.g. implantable cardioverter-defibrillator);
* Patients with any electronic/magnetic/mechanically controlled devices (e.g. sacral nerve stimulators, bladder stimulators);
* Patients with dysphagia, odynophagia or known swallowing disorder;
* Patients with known Zenker's diverticulum;
* Patients with suspected bowel obstruction or bowel perforation;
* Patients with prior bowel obstruction;
* Patients with gastroparesis or known gastric outlet obstruction;
* Patients with known Crohn's disease;
* Patients who are taking daily non-steroidal anti-inflammatory drugs (excluding prophylactic doses of aspirin) for more than six months;
* Patients who have received abdominopelvic radiotherapy treatment;
* Patients with a history of GI tract surgery (Billroth I, Billroth II, Oesophagectomy, gastrectomy or bariatric procedure);
* Patients who are pregnant or lactating;
* Patients with altered mental status that would limit their ability to swallow;
* Patients with allergy to conscious sedation, polyethylene glycol or metoclopramide;
* Patients unwilling to swallow the capsule;
* Patients with known dementia affecting ability to consent;
* Patients who have warning signs in recent years including abnormal weight loss(>10% in recent 3 month), bloody stool (except hemorrhoids), infection, etc.;
* Other inappropriate situations determined by physicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with the increasing of SCBMs during treatment period≥1 | Up to 6 weeks
  Based on diary card, researchers knew the total times of SCBMs during treatment period. The number divided by the treatment days and multiplied by 7 were the mean SCBMs per week in treatment period. Researcher compared the mean SCBMs per week with SCBMs in baseline period. "Spontaneous" suggested that no laxatives and enema were taken within 24 hours before defecation.

SECONDARY OUTCOMES:
Increase of SCBMs from baseline to treatment period | Up to 6 weeks
  Based on diary card, researchers knew the SCBMs per week during treatment period. Researchers compared them with SCBMs in baseline period.
The proportion of patients with the increasing of SCBMs ≥1 in at least 4 weeks | Up to 6 weeks
  Based on diary card, researchers knew the SCBMs of each week. We compared them with SCBMs in baseline period.
Increase of SBMs from baseline to treatment period | Up to 6 weeks
  SBM means spontaneous bowel movement.
Increase of PAC-QOL score from baseline to treatment period | Up to 6 weeks
  The PAC-QOLquestionnaire contains 28 items grouped into 4 subscales (Values, 2005) covering: Worries and concerns (11 items), Physical discomfort (4 items), Psychosocial discomfort (8 items), and Satisfaction of treatment (5 items).
  A 5-point Likert response scale, ranging from 0 (Not at all / none of the time) to 4 (Extremely / All of the time), is used over a 2-week run in period and 6-week treatment period.
The proportion of patients with the increasing of PAC-QOL score during treatment period≥1 | Up to 6 weeks
  At each visit, patients were asked to fill the PAC -QOL questionnaire. The score of PAC-QOL questionnaire in 6-week treatment period were the mean score of three times.
The proportion of patients with the increasing of PAC-SYM score during treatment period≥1 | Up to 6 weeks
  The Patient Assessment of Constipation-Symptoms (PAC-SYM) questionnaire contained 12 items ( Frank, 1999) assigned to 3 subscales: stool symptoms, rectal symptoms, and abdominal symptoms. Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe'). The lower the total score, the lower the symptom burden.
Bristol Score during treatment period | Up to 6 weeks
  Stool consistency score using Bristol Stool Form Scale (median, range)-1 for hard lumps to 7 for watery stools.
Incidence of adverse events | Up to 8 weeks
  The safety were assessed by the adverse events occured during this study.

CONTACTS AND LOCATIONS:
Overall Officials: Liao Zhuan, MD, Study Chair — Department of Gastroenterology, Changhai Hospital, the Naval Medical University
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Suares NC, Ford AC. Prevalence of, and risk factors for, chronic idiopathic constipation in the community: systematic review and meta-analysis. Am J Gastroenterol. 2011 Sep;106(9):1582-91; quiz 1581, 1592. doi: 10.1038/ajg.2011.164. Epub 2011 May 24. PMID 21606976
- [Background] Ron Y, Halpern Z, Safadi R, Dickman R, Dekel R, Sperber AD. Safety and efficacy of the vibrating capsule, an innovative non-pharmacological treatment modality for chronic constipation. Neurogastroenterol Motil. 2015 Jan;27(1):99-104. doi: 10.1111/nmo.12485. Epub 2014 Dec 6. PMID 25484196
- [Background] Nelson AD, Camilleri M, Acosta A, Boldingh A, Busciglio I, Burton D, Ryks M, Zinsmeister AR. A single-center, prospective, double-blind, sham-controlled, randomized study of the effect of a vibrating capsule on colonic transit in patients with chronic constipation. Neurogastroenterol Motil. 2017 Jul;29(7). doi: 10.1111/nmo.13034. Epub 2017 Feb 8. PMID 28177172
- [Background] Yu J, Qian YY, He CH, Zhu SG, Zhao AJ, Zhu QQ, Shao CW, Wang TG, Wang Y, Ding GL, Liao Z, Li ZS. Safety and Efficacy of a New Smartphone-controlled Vibrating Capsule on Defecation in Beagles. Sci Rep. 2017 Jun 6;7(1):2841. doi: 10.1038/s41598-017-02844-4. PMID 28588191
- [Background] Nee J, Sugarman MA, Ballou S, Katon J, Rangan V, Singh P, Zubiago J, Kaptchuk TJ, Lembo A. Placebo Response in Chronic Idiopathic Constipation: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2019 Dec;114(12):1838-1846. doi: 10.14309/ajg.0000000000000399. PMID 31592782
- [Derived] Zhu JH, Qian YY, Pan J, He C, Lan Y, Chen WN, Wang BM, Zhao W, Li JN, Li XQ, Lv B, Fan YH, Zuo XL, Li Z, Zou DW, Li ZS, Liao Z. Efficacy and safety of vibrating capsule for functional constipation (VICONS): A randomised, double-blind, placebo-controlled, multicenter trial. EClinicalMedicine. 2022 Apr 25;47:101407. doi: 10.1016/j.eclinm.2022.101407. eCollection 2022 May. PMID 35518121